CLINICAL TRIAL: NCT06218069
Title: Immuno-pet IMaging ResPonses AdministeRed Immune CheckpoiNt InhibiTor (IMPRINT)
Brief Title: Immuno-pet IMaging ResPonses AdministeRed Immune CheckpoiNt InhibiTor
Acronym: IMPRINT
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Pfizer (Industry); ImaginAb, Inc. (Industry); University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMAGIO-IMPRINT
Record Dates: First submitted 2023-12-19; First posted 2024-01-23 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: NSCLC
Keywords: neo-adjuvant; immune therapy; in vivo imaging; PETscan; anti-PD1

STUDY DESIGN:
Intervention Model Description: Arm 1: n=10 patients, who will receive a single subcutaneous injection with sasanlimab at 4-5 weeks prior to surgery.
  Arm 2: n=10 patients, who will receive a single subcutaneous injection with sasanlimab at 4-5 weeks prior to surgery, and a single dose radiation therapy in the week following sasanlimab injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Site EKUT (Tuebingen) (Active Comparator): Patients will receive a single subcutaneous administration of the immunotherapy sasanlimab in a fixed dose of 300 mg in a neo-adjuvant setting, followed by curative-intended surgery.
  Patients will also receive a radiolabeled imaging tracer [89Zr]Zr-crefmirlimab berdoxam that entails two intravenous administrations of a fixed dose of 1.5 mg protein dose labelled with activity dose 37 MBq Zirconium-89; one at baseline and one at 2 weeks after sasanlimab injection.
  Interventions: Drug: Sasanlimab; Drug: [89Zr]Zr-crefmirlimab berdoxam
- Site Radboudumc (Nijmegen) (Active Comparator): Patients will receive a single subcutaneous administration of the immunotherapy sasanlimab in a fixed dose of 300 mg in a neo-adjuvant setting, and 3 days of non-ablative dose radiation therapy starting with sasanlimab injection. This is followed by curative-intended surgery.
  Patients will also receive a radiolabeled imaging tracer [89Zr]Zr-crefmirlimab berdoxam that entails two intravenous administrations of a fixed dose of 1.5 mg protein dose labelled with activity dose 37 MBq Zirconium-89; one at baseline and one at 2 weeks after sasanlimab injection.
  Interventions: Drug: Sasanlimab; Radiation: non-ablative radiotherapy; Drug: [89Zr]Zr-crefmirlimab berdoxam

INTERVENTIONS:
Drug: Sasanlimab — 6 mL of the study drug will be administered subcutaneous injection in the abdominal fat fold. If SC injections in the abdominal location are not possible, SC injections can be administered in a distributed manner in the thighs. SC injections in the upper extremities (eg, deltoid, upper and lower arm) are not permitted. Any observed abnormality at the injection site (e.g. erythema, induration, ecchymosis, injection site pain, injection site pruritus) will be monitored and judged by the investigator to determine whether a corresponding AE should be reported.
  Other Names: humanized hinge region-stabilized IgG4 monoclonal anti-PD1 antibody; PF-06801591
Radiation: non-ablative radiotherapy — Patients will receive a total dose of 24Gy irradiation to the tumor, fractionated in 3 doses of 8Gy, on three consecutive days and starting on the day of first sasanlimab administration.
  Arms: Site Radboudumc (Nijmegen)
Drug: [89Zr]Zr-crefmirlimab berdoxam — Prior to sasanlimab injection and prior to surgery, [89Zr]Zr-crefmirlimab berdoxam (1.5 mg protein dose labelled with activity dose 37 MBq Zirconium-89) will be administered via an intravenous catheter. After 21-27 hours after injection patient will undergo a whole-body PETscan te detect CD8+ T-cell infiltration.

SUMMARY:
This study investigates whether a single subcutaneous administration of anti-PD-1 antibody can induce CD8+ T-cell tumor-infiltration that can be non-invasively monitored with [89Zr]crefmirlimab berdoxam PET imaging as an imaging biomarker.

DETAILED DESCRIPTION:
This is a two-armed open-label feasibility study with exploratory endpoints, where subjects are participating for 2 years after completement of enrollment to determine disease-free survival rates. The therapeutic intervention is a single subcutaneous administration of the humanized hinge region-stabilized IgG4 monoclonal anti-PD1 antibody PF-06801591 (sasanlimab) in a fixed dose of 300 mg in a neo-adjuvant setting, with or without radiation therapy, followed by curative-intended surgery. The diagnostic intervention is a radiolabeled imaging tracer [89Zr]Zr-crefmirlimab berdoxam that entails two intravenous administrations of a fixed dose of 1.5 mg protein dose labelled with activity dose 37 MBq Zirconium-89; one at baseline and one at 2 weeks after sasanlimab injection, to visualize CD8+ T-cells in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years
* Histologically or cytologically proven adenocarcinoma or squamous cell lung cancer
* Primary tumors >1 cm and </= 5 cm largest diameter
* Scheduled for curative surgery
* Informed consent
* Adequate bone marrow function (ANC >/= 1500, platelets >/=100k, Hgb > 9), renal function (CLCr >30 mL/min), liver function (TotalBili </= 1.5 x ULN; AST and ALT </=2.5 x ULN).

Exclusion Criteria:

* Inability to undergo SPECT or PET scans
* Pleiomorphic, lepidic, mucinous or large cell neuro-endocrine histological subtypes of non-small cell lung carcinoma
* Histologically confirmed druggable mutation (EGFR, RET, ROS, ALK, BRAF V600, NTRK, NRG1, MET ex14Sk)
* Pregnancy or lactation
* Active infection, auto-immune disease, prior organ-transplantation or haematological condition that requires medication that potentially interferes with immune cell activation.
* Documented medical history of auto-immune disease, organ-transplantation or haematological condition that potentially interferes with immune cell behavior
* Prior radiation therapy to the chest
* Splenectomy
* Enrolled in a current investigational drug trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with successful completion of curative surgery within 42 days after start of subcutaneous sasanlimab as neo-adjuvant treatment. | 2 years
  Feasibility will be determined on all patients who have entered the treatment phase of the study, i.e. received at least one course of neo-adjuvant sasanlimab. Feasibility is defined as successful completion of curative surgery within 42 days after start of neo-adjuvant treatment (= day 1). No delays will be allowed. Results will be reported in a descriptive fashion, including percentages, mean and standard deviation, median and range for the time-related measures.
The number of CTC grade ≥3 toxicity related to subcutaneous sasanlimab as neo-adjuvant treatment. | 2 years
  Safety will be defined as the number of CTC grade ≥3 toxicity related to neo-adjuvant sasanlimab. Results will be reported in a descriptive fashion.
Detection of treatment induced immune related responses after subcutaneous sasanlimab as neo-adjuvant treatment. | 2 years
  Efficacy will be defined as the detection of treatment induced immune related responses in >15% of the patients. Results will be reported in a descriptive fashion, for both cohorts of each n=10 patients (sasanlimab with and without radiotherapy).

SECONDARY OUTCOMES:
Demonstrate induction of CD8+ T-cells | 2 years
  Determine changes from baseline in immune profiles, including maturation stages, activation markers, chemokine receptors and functional markers on different lymphocyte (sub-)populations assessed by multipanel flowcytometry on samples obtained at 3 weeks and expressed in percentages and absolute numbers per mL.
Framework for PETscan interpretation | 2 years
  Determine the (changes in) relative distributions of tracer uptake (e.g., CD8+ T-cell distributions) across tumor, tumor-draining lymph node(s), spleen, bone marrow, blood pool and distant lymph nodes computed from [89Zr]Zr-crefmirlimab berdoxam PET images.
  Correlative analyses of CD8+ T-cell profiles will be done in peripheral blood at the time point of scanning and resected tumor sections.
Identify immune signatures | 2 years
  The absolute number, mean and maximum density of CD8+ T-cells/mm^2 tumor tissue will be determined and correlated with conventional pathological response assessment and clinical endpoint of 1- and 2-year recurrence free survival.
  The absolute number, mean and maximum density of other immune cell (sub-)populations will be determined by multipanel immunohistochemistry and immunofluorescence analyses on the resected tumor tissue and correlated to pathological and clinical response, as above.
Explore pathological response rate | 2 years
  The conventional pathological response assessment will be compared for both study arms and reported as absolute number and percentage of total subjects who received sasanlimab prior to surgery in that study arm.
  Comparative and descriptive analyses of immune cell signatures in peripheral blood, [89Zr]Zr-crefmirlimab berdoxam and resected tumor specimen with respect to both study arms will be performed to explore potential effect of radiotherapy on immune responses.

CONTACTS AND LOCATIONS:
Overall Officials: Michel M van den Heuvel, Prof.dr., Principal Investigator — Radboud University Medical Center (Radboudumc); Dominik Sonanini, Dr., Principal Investigator — Eberhard Karls Universitaet Tuebingen (EKUT)
Locations (2):
- Eberhard Karls Universitaet Tuebingen (EKUT), Tübingen, Germany
- Radboud University Medical Center (Radboudumc), Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Raw and/or processed data will be made available for researchers upon reasonable request.

REFERENCES:
- [Background] Rosner S, Reuss JE, Zahurak M, Zhang J, Zeng Z, Taube J, Anagnostou V, Smith KN, Riemer J, Illei PB, Broderick SR, Jones DR, Topalian SL, Pardoll DM, Brahmer JR, Chaft JE, Forde PM. Five-Year Clinical Outcomes after Neoadjuvant Nivolumab in Resectable Non-Small Cell Lung Cancer. Clin Cancer Res. 2023 Feb 16;29(4):705-710. doi: 10.1158/1078-0432.CCR-22-2994. PMID 36794455
- [Background] Reuss JE, Anagnostou V, Cottrell TR, Smith KN, Verde F, Zahurak M, Lanis M, Murray JC, Chan HY, McCarthy C, Wang D, White JR, Yang S, Battafarano R, Broderick S, Bush E, Brock M, Ha J, Jones D, Merghoub T, Taube J, Velculescu VE, Rosner G, Illei P, Pardoll DM, Topalian S, Naidoo J, Levy B, Hellmann M, Brahmer JR, Chaft JE, Forde PM. Neoadjuvant nivolumab plus ipilimumab in resectable non-small cell lung cancer. J Immunother Cancer. 2020 Sep;8(2):e001282. doi: 10.1136/jitc-2020-001282. PMID 32929052
- [Background] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N; CheckMate 816 Investigators. Neoadjuvant Nivolumab plus Chemotherapy in Resectable Lung Cancer. N Engl J Med. 2022 May 26;386(21):1973-1985. doi: 10.1056/NEJMoa2202170. Epub 2022 Apr 11. PMID 35403841
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Wakelee H, Liberman M, Kato T, Tsuboi M, Lee SH, Gao S, Chen KN, Dooms C, Majem M, Eigendorff E, Martinengo GL, Bylicki O, Rodriguez-Abreu D, Chaft JE, Novello S, Yang J, Keller SM, Samkari A, Spicer JD; KEYNOTE-671 Investigators. Perioperative Pembrolizumab for Early-Stage Non-Small-Cell Lung Cancer. N Engl J Med. 2023 Aug 10;389(6):491-503. doi: 10.1056/NEJMoa2302983. Epub 2023 Jun 3. PMID 37272513
- [Background] Cascone T, William WN Jr, Weissferdt A, Leung CH, Lin HY, Pataer A, Godoy MCB, Carter BW, Federico L, Reuben A, Khan MAW, Dejima H, Francisco-Cruz A, Parra ER, Solis LM, Fujimoto J, Tran HT, Kalhor N, Fossella FV, Mott FE, Tsao AS, Blumenschein G Jr, Le X, Zhang J, Skoulidis F, Kurie JM, Altan M, Lu C, Glisson BS, Byers LA, Elamin YY, Mehran RJ, Rice DC, Walsh GL, Hofstetter WL, Roth JA, Antonoff MB, Kadara H, Haymaker C, Bernatchez C, Ajami NJ, Jenq RR, Sharma P, Allison JP, Futreal A, Wargo JA, Wistuba II, Swisher SG, Lee JJ, Gibbons DL, Vaporciyan AA, Heymach JV, Sepesi B. Neoadjuvant nivolumab or nivolumab plus ipilimumab in operable non-small cell lung cancer: the phase 2 randomized NEOSTAR trial. Nat Med. 2021 Mar;27(3):504-514. doi: 10.1038/s41591-020-01224-2. Epub 2021 Feb 18. PMID 33603241
- [Background] Altorki NK, McGraw TE, Borczuk AC, Saxena A, Port JL, Stiles BM, Lee BE, Sanfilippo NJ, Scheff RJ, Pua BB, Gruden JF, Christos PJ, Spinelli C, Gakuria J, Uppal M, Binder B, Elemento O, Ballman KV, Formenti SC. Neoadjuvant durvalumab with or without stereotactic body radiotherapy in patients with early-stage non-small-cell lung cancer: a single-centre, randomised phase 2 trial. Lancet Oncol. 2021 Jun;22(6):824-835. doi: 10.1016/S1470-2045(21)00149-2. Epub 2021 May 18. PMID 34015311
- [Background] Cytlak UM, Dyer DP, Honeychurch J, Williams KJ, Travis MA, Illidge TM. Immunomodulation by radiotherapy in tumour control and normal tissue toxicity. Nat Rev Immunol. 2022 Feb;22(2):124-138. doi: 10.1038/s41577-021-00568-1. Epub 2021 Jul 1. PMID 34211187
- [Background] Rodriguez-Ruiz ME, Vanpouille-Box C, Melero I, Formenti SC, Demaria S. Immunological Mechanisms Responsible for Radiation-Induced Abscopal Effect. Trends Immunol. 2018 Aug;39(8):644-655. doi: 10.1016/j.it.2018.06.001. Epub 2018 Jul 11. PMID 30001871
- [Background] Hu-Lieskovan S, Braiteh F, Grilley-Olson JE, Wang X, Forgie A, Bonato V, Jacobs IA, Chou J, Johnson ML. Association of Tumor Mutational Burden and Immune Gene Expression with Response to PD-1 Blockade by Sasanlimab Across Tumor Types and Routes of Administration. Target Oncol. 2021 Nov;16(6):773-787. doi: 10.1007/s11523-021-00833-2. Epub 2021 Oct 25. PMID 34694529
- [Background] Al-Khami AA, Youssef S, Abdiche Y, Nguyen H, Chou J, Kimberlin CR, Chin SM, Kamperschroer C, Jessen B, Kern B, Budimir N, Dillon CP, Xu A, Clark JD, Chou J, Kraynov E, Rajpal A, Lin JC, Salek-Ardakani S. Pharmacologic Properties and Preclinical Activity of Sasanlimab, A High-affinity Engineered Anti-Human PD-1 Antibody. Mol Cancer Ther. 2020 Oct;19(10):2105-2116. doi: 10.1158/1535-7163.MCT-20-0093. Epub 2020 Aug 26. PMID 32847983